CLINICAL TRIAL: NCT00578357
Title: A Personalized Feedback Intervention for Problem Gamblers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Dr. John Cunningham, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 212/2007
Record Dates: First submitted 2007-12-18; First posted 2007-12-21 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Problem Gambling
Keywords: problem gambling; personalized feedback; gambling addiction
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): immediate intervention
  Interventions: Behavioral: personalized feedback intervention
- 2 (No Intervention): note: participants in this arm will receive the intervention after the 6-month follow-up (serving as control during the trial)

INTERVENTIONS:
Behavioral: personalized feedback intervention — personalized feedback will be sent to participants after they complete and return self-help materials/questionnaires
  Arms: 1

SUMMARY:
The main aim of this randomized controlled trial is to evaluate the sustained efficacy of a personalized feedback intervention for problem gamblers. Adult problem gamblers who express an interest in self-help materials for gamblers will be recruited from respondents to a random digit telephone survey, which also collects the baseline data. Subjects will be randomly assigned to receive personalized feedback about their gambling, or to a waiting list control group.

Three-month, six-month, and 12-month follow-up surveys will be conducted by mail to assess gambling over the intervening periods. Collaterals will be requested as part of the 12-month follow-up and interviewed by telephone. Gambling at three- six- and 12-months will be compared between the groups. Change in perception of gambling norms and sex will be tested as mediational and moderating variables.

DETAILED DESCRIPTION:
Most problem gamblers don't access treatment, often because of stigma, embarrassment or a desire to handle their problems on their own. However, research has demonstrated the effectiveness of self-help interventions for gambling problems, and this area deserves more attention because it addresses a cost-effective means of helping problem gamblers without requiring them to come to treatment. One promising self-help intervention for problem gamblers is personalized feedback. Such interventions have shown consistently positive results with other addictive behaviours, and our pilot test of personalized feedback materials for gamblers showed positive results. This randomized controlled study will evaluate the sustained efficacy of a personalized feedback intervention for problem gamblers in the general population of Ontario. It will also allow testing of the hypothesis that change in perception of gambling norms is a mediator in this process.

Hypothesis 1: Problem gamblers who receive the personalized feedback intervention will reduce their gambling more than problem gamblers who do not receive any intervention (waiting list control condition) by a six-month follow-up.Hypothesis 2: The effect of the intervention will be sustained through the 12-month follow-up.Hypothesis 3 (mediator hypothesis): Respondents in the intervention condition who report greater reductions in their estimates about how much others gamble between baseline and three-month follow-up will demonstrate more improvement in gambling outcomes at six-month follow-up, compared to respondents in the intervention condition who report smaller reductions in their perceived gambling norms.

The design of this study is a randomized (modified) waiting list controlled study. Subjects will be recruited via a random digit dialing telephone screener of the Ontario population. Respondents who are identified by the screener as problem gamblers and who indicate an interest in receiving, at some time in the future, a free computerized summary comparing their gambling to that of other Canadians, will be asked if they will take part in a study to "help us develop and evaluate self-help materials for gamblers." They will be told that the materials and the three-, six- and 12-month follow-up surveys would be mailed to them. Compensation is provided for the completion of each survey.

Provision of name and address will constitute consent. Subjects will be randomly assigned to condition - those in the intervention condition will be sent their personalized feedback - those in the control condition will be asked to tell us what they think should be included in self-help materials for gamblers. (Control subjects will receive the personalized feedback after the six-month follow-up.)

3-month, 6-month, and 12-month follow-up questionnaires will be sent to all subjects.

On the 12-month follow-up subjects will be asked to provide the name, address and telephone number of a collateral.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* encompassing the full range of potential problems from moderate problem gambling to gambling dependence as defined by the Canadian Problem Gambling Index (CPGI score of 3 or more)
* spent at least $100.00 in the past year on gambling
* will indicate an interest in self-help materials for problem gamblers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2007-12; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
mean number of dollars lost per month | 1 month
mean number of gambled days per month | 1 month
greatest dollar amount gambled on any day | 1 day
total CGPI score | intermittent

CONTACTS AND LOCATIONS:
Overall Officials: John Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cunningham JA, Hodgins DC, Toneatto T, Murphy M. A randomized controlled trial of a personalized feedback intervention for problem gamblers. PLoS One. 2012;7(2):e31586. doi: 10.1371/journal.pone.0031586. Epub 2012 Feb 14. PMID 22348112